CLINICAL TRIAL: NCT00107354
Title: Phase I Study of Adoptive Immunotherapy With CD8 Minor Histocompatibility (H) Antigen-Specific CTL Clones for Patients With Relapsed of AML or ALL After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Cellular Adoptive Immunotherapy in Treating Patients With Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Myelodysplastic Syndromes That Relapsed After Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 1334.00; CDR0000407784
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; T-cell adult acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Congenital Abnormalities | interventions — aldesleukin; Cytarabine; Etoposide; Mitoxantrone; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic allogeneic lymphocytes
Biological: therapeutic autologous lymphocytes
Drug: cytarabine
Drug: etoposide
Drug: mitoxantrone hydrochloride
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Biological therapies, such as cellular adoptive immunotherapy, stimulate the immune system in different ways and stop cancer cells from growing.

PURPOSE: This phase I trial is studying the side effects of cellular adoptive immunotherapy in treating patients with acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndromes that relapsed after donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxic effects of adoptive immunotherapy comprising CD8-positive minor histocompatability antigen-specific cytotoxic T-lymphocytes in patients with acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndromes that relapsed after allogeneic hematopoietic stem cell transplantation.

Secondary

* Determine the persistence of adoptively transfused T cells in vivo and assess their migration to the bone marrow in these patients.
* Determine the anti-leukemic activity of this therapy in these patients.

OUTLINE: This is a pilot, open-label, nonrandomized study.

* Leukapheresis: Patients undergo leukapheresis to obtain peripheral blood mononuclear cells (PBMCs) before transplantation. Donors undergo leukapheresis to obtain PBMCs to use as feeder cells for generating adoptive immunotherapy. Patient PBMCs are combined with donor PBMCs and expanded in vitro to generate CD8-positive minor histocompatability antigen-specific cytotoxic T-lymphocytes (CTLs) for adoptive immunotherapy.
* Transplantation: Patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation. Patients with a morphologic or flow cytometric relapse on or after day 100 post-transplantation proceed to cytoreductive chemotherapy. Patients with a molecular or cytogenetic relapse on or after day 100 post-transplantation proceed directly to adoptive immunotherapy. Patients with relapsed disease before day 100 post-transplantation are eligible to receive adoptive immunotherapy at a later date provided the patient continues to relapse and CTLs are available.
* Cytoreductive chemotherapy: The chemotherapy regimen for each patient is determined after consideration of prior chemotherapy, type of leukemia, and other clinical parameters. Two regimens to consider are:

  * Mitoxantrone IV and etoposide IV on days -6 to -2
  * High-dose cytarabine IV over 2 hours twice daily on days -6, -4, and -2 Patients achieving a complete remission after completion of cytoreductive chemotherapy proceed to adoptive immunotherapy.
* Adoptive immunotherapy: Within 2-3 days after completion of cytoreductive chemotherapy, patients receive CTLs IV over 1-2 hours on days 0, 4, 11, 21, and 28 in the absence of unacceptable toxicity. Patients with evidence of persistent disease on or after day 35 OR relapsed disease after an initial response to CTLs receive a sixth infusion of CTLs followed, no more than 24 hours later, by interleukin-2 subcutaneously once daily for up 14 total doses in the absence of unacceptable toxicity. Patients with subsequent relapsed disease after day 48 may be eligible for retreatment.

After completion of study treatment, patients are followed with bone marrow aspiration every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 25-30 patients (10-15 with acute myeloid leukemia or myelodysplastic syndromes AND 10-15 with acute lymphoblastic leukemia) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing allogeneic hematopoietic stem cell transplantation* from a major histocompatability complex (MHC)-identical related donor for 1 of the following:

  * Primary refractory acute myelogenous leukemia (AML) or acute lymphoblastic leukemia (ALL)
  * AML or ALL beyond first remission
  * Therapy-related AML at any stage
  * Philadelphia chromosome (bcr-abl)-positive p190-positive ALL at any stage
  * Acute leukemia at any stage arising from myelodysplastic syndromes or myeloproliferative disorders, including any of the following:

    * Chronic myelomonocytic leukemia
    * Chronic myelogenous leukemia
    * Polycythemia vera
    * Essential thrombocytosis
    * Agnogenic myeloid metaplasia with myelofibrosis
  * Refractory anemia with excess blasts
  * Refractory anemia with excess blasts in transformation NOTE: *Patients must be enrolled on study prior to undergoing transplantation
* Relapsed disease post-transplantation, as evidenced by 1 of the following criteria:

  * Morphologic relapse, as defined by 1 or more of the following:

    * Peripheral blasts in the absence of growth factor therapy
    * Bone marrow blasts > 5% of nucleated cells
    * Extramedullary chloroma or granulocytic sarcoma
  * Flow cytometric relapse, as defined by the appearance of cells with abnormal immunophenotype consistent with leukemia relapse in the peripheral blood or bone marrow (detected before transplantation)
  * Cytogenetic relapse, as defined by the appearance in 1 or more metaphases from bone marrow or peripheral blood cells of either a non-constitutional cytogenetic abnormality detected in at least 1 cytogenetic study performed before transplantation OR a new abnormality known to be associated with leukemia
  * Molecular relapse, as defined by 1 of the following:

    * 1 or more positive polymerase chain reaction (PCR) assays for clonotypic immunoglobulin heavy chain or T-cell receptor gene rearrangement in patients transplanted for B- or T-cell ALL respectively
    * 1 or more positive post-transplantation reverse transcription PCR assays for p190 BCR-ABL mRNA fusion transcripts in patients transplanted for Philadelphia chromosome-positive p190-positive ALL
* No grade III or IV acute graft-versus-host disease (GVHD)**
* No extensive chronic GVHD** NOTE: **At time of post-transplant relapse

PATIENT CHARACTERISTICS:

Age

* 14 and over (patients < 14 years of age may be eligible if they are deemed to be of sufficient height and weight by the pediatric attending physician)

Performance status

* Karnofsky 60-100% (at time of post-transplant relapse)

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No preexisting major nonhematopoietic organ toxicity ≥ grade 3 (at time of post-transplant relapse)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent immunosuppressive steroid therapy for GVHD allowed provided both of the following are true:

  * Able to taper steroid dose to < 0.5 mg/kg/day
  * No increase of > 1 grade in acute GVHD OR progression of chronic GVHD within 14 days after dose change

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-12; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Toxicity

SECONDARY OUTCOMES:
In vivo persistence of adoptively transferred T cells
Migration of adoptively transferred T cells to the bone marrow
Antileukemic activity

CONTACTS AND LOCATIONS:
Overall Officials: Edus H. Warren, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Warren EH, Fujii N, Akatsuka Y, Chaney CN, Mito JK, Loeb KR, Gooley TA, Brown ML, Koo KK, Rosinski KV, Ogawa S, Matsubara A, Appelbaum FR, Riddell SR. Therapy of relapsed leukemia after allogeneic hematopoietic cell transplantation with T cells specific for minor histocompatibility antigens. Blood. 2010 May 13;115(19):3869-78. doi: 10.1182/blood-2009-10-248997. Epub 2010 Jan 13. PMID 20071660
- [Derived] Rosinski KV, Fujii N, Mito JK, Koo KK, Xuereb SM, Sala-Torra O, Gibbs JS, Radich JP, Akatsuka Y, Van den Eynde BJ, Riddell SR, Warren EH. DDX3Y encodes a class I MHC-restricted H-Y antigen that is expressed in leukemic stem cells. Blood. 2008 May 1;111(9):4817-26. doi: 10.1182/blood-2007-06-096313. Epub 2008 Feb 25. PMID 18299450